CLINICAL TRIAL: NCT06839170
Title: A Multi-stage Evaluation Foundation Model for Inherited Retinal Diseases Care Needs: A Randomized Control Trial
Brief Title: An Assistant Model for IRD Care Needs: A Randomized Control Trial
Acronym: IRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EyeFM-IRDs; 2022YFC2502800 (Other Grant/Funding Number: National Key R & D Program of China)
Record Dates: First submitted 2025-02-11; First posted 2025-02-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Inherited Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retina4IRD(also designated as FM-IRDs) assisted arm (Experimental): Arm A: In the diagnostic process of IRD, retinal specialists make diagnostic decision with the assistance of FM-IRDs.
  Interventions: Other: FM-IRDs assisted
- specialist-only without AI assisted arm (Active Comparator): Arm B: In the diagnostic process of IRD, retinal specialists make independent decision-making without the assistance of FM-IRDs.

INTERVENTIONS:
Other: FM-IRDs assisted — A Foundation Model for Assisting the precision Diagnosis of Inherited Retinal Diseases: FM-IRDs
  Arms: Retina4IRD(also designated as FM-IRDs) assisted arm
Other: without FM-IRDs — without FM-IRDs

SUMMARY:
we present FM-IRD（also designated as Retina4IRD）, the first foundation model-based AI system specifically designed for genotype diagnosis of IRD by emulating clinician decision-making reasoning process. Retina4IRD is capable of processing multimodal input including color fundus photography (CFP), optical coherence tomography (OCT), and descriptive medical metadata. Trained and validated on genetically confirmed cases from centers across China, South Korea, and Poland, the system generates a ranked list of candidate pathogenic genetic variants. Retina4IRD also can generated attention heatmaps to enhance decision-making interpretability. To validate its clinical impact, we conducted a prospective multicenter RCT involving 295 participants, rigorously assessing Retina4IRD's diagnostic accuracy and real-world utility. This will improve the standardized diagnosis of IRD diseases, effectively transforming the traditional time-consuming and resource-intensive diagnostic pathway into an efficient intelligent workflow

DETAILED DESCRIPTION:
A randomized, controlled validation trial was conducted to evaluate the effectiveness of Retina4IRD (also designated as FM-IRD) in clinical settings. This trail was conducted at seven centers in China with large outpatient IRDs care .

Participants were recruited from the outpatient of IRD clinics of the participating centers, or through referrals from collaborating retinal specialists. Given that genetic testing results were unavailable at enrollment, and to prioritize the model's ability to identify patients with actionable therapeutic targets, genotypes of our randomized controlled trial were categorized into 17 classes, including mutations with available gene therapies or ongoing clinical trials. All participants provided written informed consent before enrolment assessments. All participants subsequently underwent WES testing to confirm the causative genetic mutations, which served as the gold standard for IRD gene mutation diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with clinical features suggestive of suspected IRD based on the initial assessment by the physician

Exclusion Criteria:

* Refusal to undergo WES genetic testing.
* Screening for a history of intraocular surgery in both eyes within the past 6 months;
* Subjects with severe systemic diseases, intellectual developmental disorders, psychiatric illnesses, etc.
* Patient data that the investigator deems necessary to exclude.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of IRDs | 21 days
  The top-5 gene mutation prediction accuracy, which will be assessed after all participants of the study have had WES test

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, PhD, Principal Investigator — Shanhai General Hopsital
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai
  - Shanghai general hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No